CLINICAL TRIAL: NCT07132021
Title: Efficacy of Trans-auricular Vagus Nerve Stimulation on Upper Extremity Motor Recovery in Stroke Survivors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: taVNS_UpperExtremity
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: trans-auricular vagus nerve stimulation; stroke; upper extremity function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transcutaneous vagus nerve stimulation stimulation (Experimental)
  Interventions: Device: Active taVNS
- Sham transcutaneous vagus nerve stimulation stimulation (Sham Comparator)
  Interventions: Device: Sham taVNS

INTERVENTIONS:
Device: Active taVNS — Protocol uses a 25 Hz frequency with 500 μs pulse width in biphasic configuration, operating at a 1:1 duty cycle with current intensity set to the maximum tolerable level without inducing pain. The total stimulation duration is 60 minutes. The stimulation is combined with physical therapy focused on upper extremity function.
  Arms: Active transcutaneous vagus nerve stimulation stimulation
Device: Sham taVNS — Physical therapy focused on upper extremity function with masking for transcutaneous vagus nerve stimulation
  Arms: Sham transcutaneous vagus nerve stimulation stimulation

SUMMARY:
The aim of this clinical trial is to determine if trans-auricular vagus nerve stimulation (taVNS) is effective in improving upper extremity function in stroke survivors. The primary objectives include: Investigating whether taVNS improves motor function in stroke survivors. The secondary objectives include: Assessing any potential side effects associated with the method. Investigating taVNS effects on daily routine functions and spasticity Researchers will conduct a comparative analysis between taVNS and a sham procedure (which mimics the stimulation without any actual effect) to assess its effectiveness. Participants in the trial will: Undergo taVNS combined with physical therapy or a sham procedure with physical therapy daily over a two-week period.

ELIGIBILITY:
Inclusion Criteria:

Patients aged between 18 and 75 years, with motor impairment in the upper extremity caused by unilateral ischemic or hemorrhagic stroke with stroke onset within the last five years.

Exclusion Criteria:

* Patients with any contraindication to taVNS, peripheral upper extremity injuries, use of medication affecting cortical excitability in the past 3 months, use of botulinum toxin in the past 3 months, presence of any other neurological disorder, or significant cognitive deficits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Upper extremity Motor Function (Fugl-Meyer Assessment - Upper Extremity) | Baseline (Day 0), mid-intervention (day 5) and post-intervention (day 10)
  The Fugl-Meyer Assessment for Upper Extremity (FMA-UE) will be used to evaluate motor impairment and recovery of the paretic upper extremity. It consists of items from sections III and IV, assessing motor function, coordination, and speed, with a maximum score of 66 points. Higher scores indicate lower motor impairment. A minimal clinically important difference (mCID) is defined as a change (Δ) of 5 or more points between baseline and post-intervention scores.

SECONDARY OUTCOMES:
Manual Dexterity (Box and Block Test) | Baseline (Day 0), mid-intervention (day 5) and post-intervention (day 10)
  The Box and Block Test (BBT) will assess manual dexterity of the paretic upper extremity. It counts the number of wooden blocks (2.5 x 2.5 x 2.5 cm) transferred from one compartment to another over a central divider within one minute. The minimal detectable change (MDC) is defined as a difference of 5 blocks per minute.
Independence (Functional Independence Measure) | Baseline (Day 0), mid-intervention (day 5) and post-intervention (day 10)
  The Functional Independence Measure (FIM) assesses the level of independence through motor and cognitive subscales. Each item is scored from 1 to 7. Total score classifications: complete dependence (18-45), moderate independence (46-99), and complete independence (100-126). The MDC is defined as 17 points for the motor section, 3 points for the cognitive section, and 22 points for the total score.
Spasticity (Modified Ashworth Scale) | Baseline (Day 0), mid-intervention (day 5) and post-intervention (day 10)
  The Modified Ashworth Scale (MAS) will assess spasticity in finger, wrist, elbow, and shoulder flexors of the paretic upper extremity. It uses a 6-point scale (0 to 5) to quantify muscle tone. The minimal clinically important difference (mCID) is defined as a reduction of at least one point in spasticity score.
Health-Related Quality of Life (Stroke-Specific Quality of Life Scale) | Baseline (day 0), mid-intervention (day 5), post-intervention (day 10)
  The Stroke-Specific Quality of Life Scale (SS-QOL) assesses stroke-related quality of life across 12 domains, using 49 items. Scores range from 49 to 245, with higher scores indicating better quality of life. The MDC is 4.7 points for the total score, 2.1 for the physical subscore, and 2.8 for the psychosocial subscore.
Multidimensional Stroke Impact (Stroke Impact Scale) | Baseline (Day 0), mid-intervention (Day 5), post-intervention (Day 10)
  The Stroke Impact Scale (SIS) is a self-reported questionnaire assessing multiple consequences of stroke including strength, hand function, mobility, ADLs/IADLs, memory and thinking, communication, emotion, and social participation. It is designed to capture the broader impact of stroke on health and quality of life.
Global Perception of Change (Patient Global Impression of Change) | Baseline (Day 0), mid-intervention (Day 5), post-intervention (Day 10)
  The Global Perception of Change Scale (also referred to as Patient Global Impression of Change - PGIC) assesses the participant's perceived improvement at post-intervention. It includes 7 options, ranging from "no change or condition worsened" to "a great deal better, considerable improvement that made all the difference."

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Monte-Silva, PhD in Neurosciences, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No